CLINICAL TRIAL: NCT01516905
Title: PET/CT Imaging of Malignant Brain Tumors With a Novel Radioiodinated Phospholipid Ether Analogue 124I-NM404
Brief Title: PET/CT Imaging of Malignant Brain Tumors With 124I-NM404
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: RO11310; 1R01CA158800-01 (NIH); NCI-2012-02042 (Registry Identifier: NCI Trial ID); 2011-0452 (Other: Institutional Review Board); A539300 (Other: UW Madison); SMPH\RADIOLOGY\RADIOLOGY (Other: UW Madison)
Record Dates: First submitted 2012-01-10; First posted 2012-01-25 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-02

CONDITIONS: Glioblastoma; Brain Metastases
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- I124-NM404 brain metastases or GBM imaging: determining appropriate imaging timepoints. Image at 6 hour, 24 hour and 48 hour post injection of I-124NM404
  Interventions: Drug: NM404

INTERVENTIONS:
Drug: NM404 — injection of either 2.0mCi or 5.0mCi I-124 NM404
  Other Names: PET imaging with I-124 NM404

SUMMARY:
The purpose of this study is to evaluate diagnostic imaging techniques using 124I-NM404 PET/CT in humans with brain metastases and GBMs. This goal will be accomplished by determining the optimal PET/CT protocol and comparing PET tumor uptake to MRI and calculating tumor dosimetry. A future aim of this study will be to compare non-invasive PET/CT and MRI findings with pathological specimens, which is the gold standard but is invasive and impractical in many cases, to determine the sensitivity and specificity of both techniques for accurately detecting tumor infiltration. The data obtained from this study will be used to develop larger diagnostic and therapeutic trials in brain tumors. The long-term goals of this research are to improve the diagnosis and treatment of malignant brain tumors by using radioiodinated NM404.

ELIGIBILITY:
Inclusion Criteria:

1. Participants will have a contrast enhanced brain MRI which documents evidence of GBM or metastatic brain tumor
2. Tumor size at least 1.5 cm in greatest axial dimension on MRI. MRI must be obtained within 2 months of study inclusion
3. Female patients must not be pregnant or breast feeding and both women of childbearing potential, and men, must use appropriate means of contraception and must be maintained for at least 45 days after injection of I-124 NM404. Participants must not attempt to become pregnant during this time
4. Platelet count must be ≥ 160,000/µl, Hematocrit must be ≥ 22%, Leukocyte count must be ≥ 3,000/µL, Creatinine must be ≤ 2.5 mg/dL, ALT must be ≤ 130 U/L, AST must be ≤ 100 U/L, and urine or serum pregnancy test must be negative for pregnancy
5. Karnofsky score ≥ 60
6. For brain metastases patients: targeted brain therapy (radiation or drug) must have concluded ≥2 months prior to injection of 124I-NM404
7. For GBM tumors confirmed by surgical biopsy or suspected by MRI: no previous surgical resection (except for biopsy) or systemic or radiation therapy targeted to the GBM tumor -

Exclusion Criteria:

1. Life expectancy of < 3 months
2. Allergy to potassium iodide (SSKI or Thyroshield)
3. Planned surgical resection or biopsy after injection of 124I-NM404 and prior to completion of the 3rd PET/CT scan
4. Unwilling or unable to complete 3 separate PET/CT imaging sessions of 90 minutes each over 3 days -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited when seen by oncologists in the UWCCC clinic.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2011-12; Primary Completion 2016-05-17 (Actual); Study Completion 2016-05-17 (Actual)

PRIMARY OUTCOMES:
tumor to background ratios | 48hrs
  patients will be imaged at 3 different times out to 48 hrs post injection. Images will be evaluated based on tumor/background, dimensions/volumes and a qualitative score

CONTACTS AND LOCATIONS:
Overall Officials: Lance Hall, MD, Principal Investigator — University of Wisconsin, Madison; Scott Perlman, MD, MS, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/